CLINICAL TRIAL: NCT00727766
Title: Phase I Study of Oral Clofarabine Consolidation in Adults Aged 60 and Older With Acute Myeloid Leukemia
Brief Title: Oral Clofarabine for Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0853 / 201108049
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Clofarabine; Clolar; AML; Consolidation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 (Experimental): Clofarabine 1 mg for 14 days followed by 14 days of rest. Each cycle is 28 days long.
  Interventions: Drug: Clofarabine
- Cohort 2 (Experimental): Clofarabine 2 mg for 21 days followed by 7 days of rest. Each cycle is 28 days long.
  Interventions: Drug: Clofarabine
- Cohort 3 (Experimental): Clofarabine 3 mg for 21 days followed by 7 days of rest. Each cycle is 28 days long.
  Interventions: Drug: Clofarabine
- Cohort 4 (Experimental): Clofarabine 4 mg for 21 days followed by 7 days of rest. Each cycle is 28 days long.
  Interventions: Drug: Clofarabine
- Cohort 5 (Experimental): Clofarabine 5 mg for 21 days followed by 7 days of rest. Each cycle is 28 days long.
  Interventions: Drug: Clofarabine
- Cohort 6 (Experimental): Clofarabine 6 mg for 21 days followed by 7 days of rest. Each cycle is 28 days long.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine
  Other Names: Clolar

SUMMARY:
This is a phase I study designed to test the safety of oral clofarabine when given as consolidation therapy to older patients with AML in remission.

DETAILED DESCRIPTION:
The prognosis of acute myeloid leukemia (AML) in patients 60 and older is dismal with traditional therapy. Several factors contribute to the poor prognosis of older individuals, including the increased incidence of the multidrug resistance efflux pump, comorbidities and unfavorable cytogenetics. The recently reported AML-13 and ALFA trials suggest that less intense consolidation in this population is at least equivalent to more intense, induction style efforts.

Clofarabine is a next generation nucleoside analogue that was designed to optimize the favorable attributes of fludarabine and cladribine, while minimizing toxicity. The intravenous formulation has shown considerable activity in older patients with AML who have been considered either unfit for or unlikely to benefit from conventional therapy. Additionally, clofarabine has an oral formulation that patients may find more acceptable for consolidation therapy rather than multiple courses of intravenous medications, administered over several days.

This study is designed as a traditional 3x3 phase I trial with the intention of defining the maximum tolerated dose of oral clofarabine consolidation for older patients with AML in remission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Myeloid Leukemia according to WHO criteria
* Age ≥ 60 years at enrollment
* Patients must be in complete remission by bone marrow examination, within 30 days of enrollment, following treatment with a cytotoxic induction chemotherapy regimen (such as 7+3)

  * Complete remission must be confirmed by bone marrow biopsy
  * If one cycle of consolidation was administered, then patient may be within 60 days of the confirmation of complete remission by bone marrow biopsy
  * Minimum platelet count of 100,000
* Patients may have received "low-intensity" therapy (i.e. decitabine, lenalidomide, etc) prior to traditional induction chemotherapy.
* Patients may have received 1 cycle of cytarabine-based consolidation therapy.
* Patients must have an ECOG performance status of 0-2 at the beginning of consolidation therapy.
* Have adequate renal and hepatic functions as indicated by the following laboratory values:

  * Serum creatinine ≤ 1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is black)
  * Serum total bilirubin ≤ 1.5 mg/dL × upper limit of normal (ULN) except for unconjugated hyperbilirubinemia secondary Gilbert's syndrome
  * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 × ULN
  * Alkaline phosphatase ≤ 2.5 × ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide signed valid written informed consent or when appropriate, have an appointed legally authorized representative who is capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide signed valid written informed consent for the benefit of the patient.
* Male and female patients who are of child bearing potential must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.
* Patients MAY have received prior therapy with purine analogs (such as fludarabine and cladribine).

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* The diagnosis of AML-M3 (acute promyelocytic leukemia) characterized by translocations involving the retinoic acid receptor-alpha (RAR-alpha) gene.
* Use of investigational agents within 2 weeks or any anticancer therapy within 2 weeks before study entry. The patient must have recovered from all acute toxicities from any previous therapy.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Have currently active gastrointestinal disease, or prior surgery that may affect the ability of the patient to absorb oral clofarabine.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose limiting toxicity (DLT) | DLT - 1st cycle (28 days), MTD - completion of 1st cycle by all patients in all cohorts

SECONDARY OUTCOMES:
Adverse events by grade and attribution | Start of treatment through 30 days post-last dose
Disease-free survival | Every 6 months for 3 years
Overall survival | Every 6 months for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Camille N. Abboud, M.D., Principal Investigator — Washington Univerisity
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Jacoby MA, Martin MG, Uy GL, Westervelt P, Dipersio JF, Cashen A, Stockerl-Goldstein K, Vij R, Luo J, Reineck T, Bernabe N, Abboud CN. Phase I study of oral clofarabine consolidation in adults aged 60 and older with acute myeloid leukemia. Am J Hematol. 2014 May;89(5):487-92. doi: 10.1002/ajh.23663. Epub 2014 Mar 3. PMID 24415560
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu